CLINICAL TRIAL: NCT04717609
Title: Surgeon Performed Saphenous Nerve Block at the Medial Femoral Condyle for Arthroscopic Partial Meniscectomy and Meniscus Repair: A Randomized Control Trial
Brief Title: Saphenous Nerve Block for Partial Meniscectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JHOR 20D.975
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Pain, Joint; Pain, Procedural; Meniscectomy
MeSH Terms: conditions — Arthralgia; Pain, Procedural | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Partial Meniscectomy without Saphenous Nerve Block (Active Comparator): Participants scheduled for partial meniscectomy will preoperatively receive 0.5% ropivacaine with epinephrine
  Interventions: Drug: Ropivacaine injection
- Partial Meniscectomy with Saphenous Nerve Block (Experimental): Participants scheduled for a partial meniscectomy will preoperatively receive a saphenous nerve block at the medial femoral condyle in addition to an injection of 0.5% ropivacaine with epinephrine
  Interventions: Procedure: Saphenous Nerve Block; Drug: Ropivacaine injection

INTERVENTIONS:
Procedure: Saphenous Nerve Block — Preoperative Saphenous Nerve Block for partial Meniscectomy
  Arms: Partial Meniscectomy with Saphenous Nerve Block
Drug: Ropivacaine injection — preoperatively the participant will receive an injection ar the surgical site of 5 milliliters (mL) of 0.5% ropivacaine

SUMMARY:
Partial meniscectomy and meniscus repair are two of the most common orthopedic surgery procedures. As these procedures are being increasingly performed in ambulatory surgical centers, there has been a shift towards providing improved analgesia to ensure timely discharge, as well as preventing unwanted pain and side effects. As such, it has become common practice to use an intra-articular injection of local anesthetic to achieve post-operative pain control. However, these effects are short lived, requiring a multimodal approach to analgesia. To date, no optimal pain control strategy has been described for arthroscopic partial meniscectomy or meniscus repair. The purpose of this study is to examine the outcomes of subcutaneous saphenous nerve block with 0.5% ropivacaine at the medial femoral epicondyle/adductor hiatus plus portal 0.5% ropivacaine injection vs portal 0.5% ropivacaine injection alone for patients undergoing arthroscopic partial meniscectomy or meniscus repair.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Scheduled for arthroscopic meniscectomy or meniscus repair

Exclusion Criteria:

* Multiple-ligament injury
* Primary ACL reconstruction or ACL revision reconstruction
* Articular cartilage restoration surgery
* Evidence of microfracture
* History of allergy to local anesthetics
* Pre-existing saphenous neuropathy
* Unable to be prescribed opioids due to allergy or other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-01-25 (Estimated); Primary Completion 2022-01-25 (Estimated); Study Completion 2022-01-25 (Estimated)

PRIMARY OUTCOMES:
Reduced Pain Levels | 10 days
  This will be measured by Participant Opioid Use will be collected everyday for 10 days after surgery
Quality of Recovery | 20 minutes
  After surgery while in the recovery room a 40 question survey will be administered regarding your comfort level, emotional state and pain
Reduced Pain Levels | 10 days
  This will be measured using the numeric rating score (NRS). It will be collected at 1 and 10 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States